CLINICAL TRIAL: NCT02872519
Title: PET Imaging of Ovarian Carcinoma With 18F-FSPG
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marta Crispens, MD, Professor, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC GYN 15142
Record Dates: First submitted 2016-07-26; First posted 2016-08-19 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — 4-(3-fluoropropyl)glutamic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients receive (S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG) PET scans. Patients undergo PET imaging scans during 0-45 minutes, 60-75 minutes, and 105-120 minutes after injection and within 4 weeks prior to surgery (Cohort A) or within 4 weeks of SOC imaging at diagnosis and prior to subsequent treatment (Cohort B).
  Interventions: Drug: (S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG); Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: (S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG) — Given by IV
Procedure: Positron Emission Tomography — Undergo scan
Other: Laboratory Biomarker Analysis — Laboratory Biomarker Analysis

SUMMARY:
This clinical trial studies positron emission tomography (PET) imaging utilizing 18F-FSPG [(S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid], a glutamic acid derivative, to image patients with ovarian cancer before undergoing surgery or transplant. Diagnostic procedures, such as 18F-FSPG PET, may help find and diagnose ovarian cancer and find out how far the disease has spread.

ELIGIBILITY:
Inclusion Criteria:

* Have a presumed diagnosis of advanced stage epithelial ovarian, fallopian tube, or peritoneal.

  * Pelvic mass and/or omental caking with Ca-125:CEA ratio 25:1.

    * Adequate performance status, ECOG 0, 1, 2.
* Adequate organ function:

  * PCV > 30 (with or without transfusion)
  * WBC: 3000 - 10,000 The lower level of normal for total WBCs is 4,000, but the NCI considers levels of 3,000- 4,000 as mild suppression for drug trials, specifically not requiring treatment.
  * Platelet count > 150, 000 and < 1,000,000
  * Cr < 1.5
  * LFTS < 1.5 x ULN
* Have undergone or have agreed to undergo standard of care CT of the chest, abdomen, and pelvis. 18F-FSPG PET imaging will be performed as investigational studies.
* No prior treatment for ovarian cancer
* have undergone or agree to undergo standard of care imaging for ovarian cancer with CT chest, abdomen, and pelvis.

Exclusion Criteria:

* Have non-invasive or non-epithelial ovarian cancer on pathological confirmation.
* Pregnant and breastfeeding
* Poorly controlled diabetes mellitus (fasting blood glucose level > 200 mg/dL).
* Other poorly controlled medical conditions that in the opinion of the surgeon, make them not a candidate for primary cytoreductive surgery.
* CT of chest, abdomen, pelvis demonstrates:

  * Any disease in the thoracic cavity > 1 cm.
  * Any suprarenal lymphadenopathy > 1 cm.
  * Liver metastases > 1 cm.
  * Disease in the porta hepatis or gallbladder fossa > 1 cm.
  * Pleural effusion > 50% volume of the chest cavity on chest x-ray.
  * Omental extension to the stomach, spleen, or lesser sac.

    * Extension to the pelvic sidewall (this criteria may also be assessed on physical examination.
    * involvement of the root of the mesentery.
* Decline procedures that might be necessary for optimal primary cytoreduction (i.e. colostomy or splenectomy).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Lesion (S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG) PET standard uptake values | Up to 2 years
Number of lesions detected by(S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG) PET | Up to 2 years
Number of lesions detected by (S)-4-(3-[18F]Fluoropropyl)-L-glutamic acid (18F-FSPG) PET imaging before and after neoadjuvant chemotherapy treatment | Up to 2 years

SECONDARY OUTCOMES:
Immunohistochemistry evaluation of xC- and CD 44 of resected malignant ovarian cancer with a measurement of strength of staining from 0-3. | Up to 2 years
  All imaging data (SUV) will be correlated to definitive, ex vivo diagnostic pathology and immunoreactivity (xC-, CD44), which will be carried out for every patient with resected tissue. and, when IHC scoring will be in terms of strength of immunostaining (scored on an ordinal scale of 0 3). This treatment of lesion-based sensitivity and specificity has not been previously described in the ovarian cancer literature.
Proportion of patients whose surgical resection by novel imaging classification changed following validation by histological confirmation | Up to 2 years
Proportion of patients whose response to chemotherapy changed by Response Evaluation Criteria in Solid Tumors criteria | Up to 2 years
Conditional predictive models of imaging performance and agreement | Up to 2 years
  We will test that lesion 18F-FSPG PET SUV's are significantly greater than background (normal liver tissue) by tissue assessment of number of lesions noted in each arm and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Crispens, MD, Principal Investigator — Vanderbilt University Medical Center